CLINICAL TRIAL: NCT04361149
Title: Evaluation of Motor Unit Abnormalities After Experimentally Induced Sensitization Using Capsaicin: A Randomized, Double-Blinded, Placebo-Controlled Study
Brief Title: Motor Unit Abnormalities After Experimentally Induced Sensitization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Dinesh Kumbhare, Affiliate Scientist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MotorUnitsCapsaicin
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Central Sensitisation; Motor Disorders
Keywords: Central Sensitization; Surface Electromyography; Intramuscular Electromyography; Motor Unit; Recruitment
MeSH Terms: conditions — Motor Disorders | interventions — Capsaicin

STUDY DESIGN:
Intervention Model Description: A randomized placebo controlled trial using 2 treatments: 1) placebo cream 2) capsaicin cream (0.075%) (Zostrix HP)
Who Masked: Participant
Masking Description: The participants were blinded by the cream treatment given. Both creams were in a concealed, blank, container
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Placebo Topical (Placebo Comparator): The cream was a lipobase cream, applied topically to the participants upper back, on their left side.
  Interventions: Device: Delsys Trigno Galileo System; Device: Excaliber, Natus Medical; Other: Placebo Cream
- Capsaicin Topical (Active Comparator): Capsaicin Cream (0.075%), applied topically to the participants upper back, on their left side.
  Interventions: Drug: Capsaicin Topical Cream (0.075%); Device: Delsys Trigno Galileo System; Device: Excaliber, Natus Medical

INTERVENTIONS:
Drug: Capsaicin Topical Cream (0.075%) — Capsaicin cream will be administered as a topical skin cream
  Other Names: Zostrix HP
  Arms: Capsaicin Topical
Device: Delsys Trigno Galileo System — A wireless surface EMG device. The sensors will be placed on the trapezius and the infraspinatus muscle, and a recording will be performed.
Device: Excaliber, Natus Medical — Intramuscular EMG machine. The intramuscular electrode will be inserted into the trapezius and a recording will be performed.
Other: Placebo Cream — Placebo cream will be administered as a topical skin cream
  Arms: Placebo Topical

SUMMARY:
Central sensitization is a condition that represents a cascade of neurological adaptations, resulting in an amplification of nociceptive responses from noxious and non-noxious stimuli. This phenomenon presents itself in a vast majority of chronic pain syndromes. Previous evidence has shown that central sensitization results in afferent nociceptor and dorsal horn abnormalities; however, a link between whether this abnormality translates into motor output and more specifically, ventral horn abnormalities, needs to be further explored. Twenty participants were recruited and either a topical capsaicin or a placebo topical cream was applied to their back to induce a transient state of sensitization. Surface electromyography(sEMG) and intramuscular electromyography(iEMG) were used to record motor unit activity from the trapezius and infraspinatus muscles before and after application of capsaicin/placebo. Motor unit recruitment and variability were analyzed in the sEMG and iEMG respectively

DETAILED DESCRIPTION:
Central sensitization describes a state of neuronal hyper-excitability in the central nervous system that may occur due to malfunction of spinal and supraspinal pain facilitatory and inhibitory circuits resulting in amplification of somatosensorial responses. Beyond somatosensorial changes, alteration in motor function can also be present with pain, and may be a reflex of neuromuscular function impairment. A normal afferent input and normal central processing circuitry is essential to deliver normal efferent output. However, the influence of the changes that occur within the dorsal horn on the ventral horn remain largely ill defined.

Motor unit assessment is crucial in evaluating diseases and abnormalities within the ventral horn. Activity of the ventral horn, where anterior horn cells reside, is very important for motor unit activation. Surface EMG (sEMG) and intramuscular EMG (iEMG) can be used to assess the neural drive to muscles, by recording motor units to understand the effects of central sensitization on motor control and the ventral horn. Based on Henneman's size principle, motor units should be recruited in the same order, with smaller units being recruited first. This principle presents an opportunity to investigate if central sensitization creates abnormalities on the motor unit level.

Previously, central sensitization has been induced in healthy subjects to examine its neurophysiological effects via capsaicin. Capsaicin, a chilli pepper extract, can be used to effectively induce experimental transient states of central sensitization. The presence of expanded sensorial responses and the involvement of the spinal nociceptive system post capsaicin have been largely tested by means of quantitative sensory testing methods and electromyography (EMG).

Despite the usefulness of experimental capsaicin to better understand the sensorial abnormalities, its impact on motor function and motor unit recruitment are lesser studied. Evidence suggests that nociceptive input by peripheral capsaicin exerts a centrally-mediated inhibitory effect on motor function. A decrease in root mean squared (RMS) amplitude during exercise at the time of peak sensitization was measured by needle EMG. However, the effect that capsaicin-induced sensitization has on individual motor units or on their recruitment patterns has not been previously examined.

The purpose of this study was to determine whether topical capsaicin-induced sensitization has any influence on ventral horn activity. We hypothesize that capsaicin induces a change in individual motor unit activity, as well as the recruitment pattern of many motor units, and may affect motor unit activity at different segmental levels from the level of capsaicin application.

Participants:

Twenty-three healthy participants, age between 20-70 years old, with no direct trauma to cervicothoracic region within the past 30 days, no past medical history of inflammatory disorders as rheumatoid arthritis, no neurodegenerative disorders such as Parkinson's disease nor motor neurone diseases as amyotrophic lateral sclerosis, or other neuromuscular disorder were recruited for this study. Also, included subjects had a normal body mass index (18.5 - 24.9) and had a pain visual analogue scale (VAS) below 3 indicating low pain severity. Since prevalence of neck pain in the general population is high, mild pain or aches are not necessarily related to an abnormality of the underlying muscle. Participants had to be able to communicate in English. Participants were excluded if they had persistent pain for more than 3 months.

Experimental Protocol:

An initial screening was performed to assess eligibility in the study. Each participant was seated upright with their hands comfortably on their lap and asked to relax their neck and shoulder muscles. The physician member of the research team then assessed the patients' pain intensity by visual analogue scale (VAS). VAS ranges from 0 to 100 mm which 0 mm reflecting no pain at all and 100 mm representing the worst imaginable pain. Following this, brush allodynia, a clinical technique used to identify pain due to a stimulus that does not normally provoke pain, was performed to confirm presence of central sensitization. To map out borders of secondary allodynia, subjects were instructed to recognize a distinct alteration in the sensation perception such as increased burning, intense pricking, or an unpleasant sensation, and that location was marked. Brush allodynia score (BAS) was calculated as the distance between the farthest points marked on the superior and inferior axis multiplied by the distance between the farthest points marked on the medial and lateral axis as previously described by Cavallone et. al. The VAS and the presence of central sensitization by means of BAS were assessed at baseline (pre) before the induction of sensitization and twenty minutes after (post).

Upon successful screening of inclusion and exclusion criteria, participants had their left side area of skin (overlying the upper trapezius and infraspinatus muscles) cleansed with alcohol preparation pads and water. The skin was abraded with '3M Red Dot' abrasive strips before application of the surface electromyogram (Trigno Galileo sensors, Delsys Inc.). Electrodes were placed in 4 areas: the muscle belly of the upper trapezius, and the infraspinatus, as well as reference electrodes on C7 and the acromion. These electrodes were 4 channel EMG sensors and had their signals filtered from 20 - 450 Hz. The sEMG recordings were wirelessly transmitted to the Trigno base station, which relays and compiles the data to Neuromap (Delsys Inc.) for signal analysis. A monopolar needle electrode was inserted into the upper fibers of trapezius muscle and its reference was placed at the mid-clavicle point. Using this setup intramuscular recordings of single motor units were performed using an Excaliber, Natus Medical clinical electrodiagnostic machine.

Electromyograms recordings before application of intervention

Participants were instructed to perform horizontal shoulder abductions from 0° to 90° and then from 90° to 0° for 1 minute. The study subject was verbally cued to move their arm every 2 seconds. sEMGs were recorded during this time. Upon completion of this task, a monopolar intramuscular needle electrode was placed directly into the upper trapezius muscle. Participants were then instructed to gently contract their trapezius muscle by shrugging their shoulder, enough to recruit only the first motor unit in that region. Visual feedback of the signal was given to the subject to ensure that only the first motor unit was activated for the movement. The signal from this motor unit was then optimized for initial deflection from baseline and amplitude characteristics before recordings were made. iEMG recordings were recorded for 30 seconds at a sampling frequency of 6 kHz.

Application of intervention

Participants received either a dose of 2.5 ml (75µg/ml) capsaicin cream (treatment, Zostrix brand) or skin lotion (placebo) which was inert and caused no sensitization effects. Participants were also blinded to the delivered treatment, using concealed containers for the creams. The location of application was a 10 cm by 10 cm square on trapezius muscle which extended from T3 to T8 on the left side that all recordings were conducted.

After collection of the baseline sEMG and iEMG recordings, a trained medical professional applied the capsaicin / placebo cream directly to the region of skin in a standardized 10 cm x 10 cm square at the spinal levels T3-T8, to sensitize the nociceptive afferents within that region. A twenty-minute waiting period was used to enable the sensitizing effects of capsaicin to take effect.

Electromyograms recordings after application of intervention

To confirm the presence of central sensitization, brush allodynia was used to detect mechanical allodynia outside the region of the primary nociception - region of topical placement - which is the region of secondary allodynia. Upon confirmation of central sensitization, in participants with application of topical capsaicin, participants were entered into the experimental arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* subject with a normal body mass index (18.5 - 24.9)
* a pain visual analogue scale (VAS) below 3 indicating low pain severity

Exclusion Criteria:

* medical history of inflammatory disorders as rheumatoid arthritis
* neurodegenerative disorders such as Parkinson's disease
* motor neurone diseases as amyotrophic lateral sclerosis, or other neuromuscular disorder

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Pain and Presence of Central Sensitization | 3 weeks
  Visual Analogue Scale(0-no pain to 10-worst pain imaginable) will measure the amount of burning pain experienced by the intervention

SECONDARY OUTCOMES:
Motor Unit Sequence Difference | 3 months
  The recruitment order of the pre motor unit and post motor units will be examined, determining how much the recruitment order changed
Variance of Motor Unit Action Potential | 3 months
  The difference in variance within the pre recorded MUAP train and post recorded MUAP train will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Kumbahre, PhD, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The University Health Network has a high importance on patient confidentiality. For ethics approval, this was complied with these standards, upholding the patient confidentiality standard at UHN.

REFERENCES:
- [Background] Schopflocher D, Taenzer P, Jovey R. The prevalence of chronic pain in Canada. Pain Res Manag. 2011 Nov-Dec;16(6):445-50. doi: 10.1155/2011/876306. PMID 22184555
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Grossschadl F, Freidl W, Rasky E, Burkert N, Muckenhuber J, Stronegger WJ. A 35-year trend analysis for back pain in Austria: the role of obesity. PLoS One. 2014 Sep 10;9(9):e107436. doi: 10.1371/journal.pone.0107436. eCollection 2014. PMID 25207972
- [Background] Boyle JP, Honeycutt AA, Narayan KM, Hoerger TJ, Geiss LS, Chen H, Thompson TJ. Projection of diabetes burden through 2050: impact of changing demography and disease prevalence in the U.S. Diabetes Care. 2001 Nov;24(11):1936-40. doi: 10.2337/diacare.24.11.1936. PMID 11679460
- [Background] Langley PC, Ruiz-Iban MA, Molina JT, De Andres J, Castellon JR. The prevalence, correlates and treatment of pain in Spain. J Med Econ. 2011;14(3):367-80. doi: 10.3111/13696998.2011.583303. Epub 2011 May 17. PMID 21574899
- [Background] Duenas M, Salazar A, Ojeda B, Fernandez-Palacin F, Mico JA, Torres LM, Failde I. A nationwide study of chronic pain prevalence in the general spanish population: identifying clinical subgroups through cluster analysis. Pain Med. 2015 Apr;16(4):811-22. doi: 10.1111/pme.12640. Epub 2014 Dec 19. PMID 25530229
- [Background] S. D. Phillips CJ, Chronic pain: a health policy perspective.In: S. Rashiq, D. Schopflocher, P. Taenzer and E. Jonsson, Eds., Weinheim: Wiley, 2008: 41-50.
- [Background] Latremoliere A, Woolf CJ. Central sensitization: a generator of pain hypersensitivity by central neural plasticity. J Pain. 2009 Sep;10(9):895-926. doi: 10.1016/j.jpain.2009.06.012. PMID 19712899
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Sterling M, Jull G, Wright A. The effect of musculoskeletal pain on motor activity and control. J Pain. 2001 Jun;2(3):135-45. doi: 10.1054/jpai.2001.19951. PMID 14622823
- [Background] Hossain MZ, Unno S, Ando H, Masuda Y, Kitagawa J. Neuron-Glia Crosstalk and Neuropathic Pain: Involvement in the Modulation of Motor Activity in the Orofacial Region. Int J Mol Sci. 2017 Sep 26;18(10):2051. doi: 10.3390/ijms18102051. PMID 28954391
- [Background] Wallwork SB, Grabherr L, O'Connell NE, Catley MJ, Moseley GL. Defensive reflexes in people with pain - a biomarker of the need to protect? A meta-analytical systematic review. Rev Neurosci. 2017 May 24;28(4):381-396. doi: 10.1515/revneuro-2016-0057. PMID 28475100
- [Background] Henderson RD, McCombe PA. Assessment of Motor Units in Neuromuscular Disease. Neurotherapeutics. 2017 Jan;14(1):69-77. doi: 10.1007/s13311-016-0473-z. PMID 27600517
- [Background] Enoka RM. Physiological validation of the decomposition of surface EMG signals. J Electromyogr Kinesiol. 2019 Jun;46:70-83. doi: 10.1016/j.jelekin.2019.03.010. Epub 2019 Mar 21. PMID 31003192
- [Background] Merletti R, Farina D. Analysis of intramuscular electromyogram signals. Philos Trans A Math Phys Eng Sci. 2009 Jan 28;367(1887):357-68. doi: 10.1098/rsta.2008.0235. PMID 19008187
- [Background] HENNEMAN E, SOMJEN G, CARPENTER DO. FUNCTIONAL SIGNIFICANCE OF CELL SIZE IN SPINAL MOTONEURONS. J Neurophysiol. 1965 May;28:560-80. doi: 10.1152/jn.1965.28.3.560. No abstract available. PMID 14328454
- [Background] Torebjork HE, Lundberg LE, LaMotte RH. Central changes in processing of mechanoreceptive input in capsaicin-induced secondary hyperalgesia in humans. J Physiol. 1992 Mar;448:765-80. doi: 10.1113/jphysiol.1992.sp019069. PMID 1593489
- [Background] W. Willis. Central sensitization and plasticity following intense noxious stimulation. In: E. Mayer and H. Raybould, Eds. Basic and clinic aspect of chronic abdominal pain. New York, NY: Elsevier, 1993: 201-207.
- [Background] Willis WD. Role of neurotransmitters in sensitization of pain responses. Ann N Y Acad Sci. 2001 Mar;933:142-56. doi: 10.1111/j.1749-6632.2001.tb05821.x. PMID 12000017
- [Background] Frymoyer AR, Rowbotham MC, Petersen KL. Placebo-controlled comparison of a morphine/dextromethorphan combination with morphine on experimental pain and hyperalgesia in healthy volunteers. J Pain. 2007 Jan;8(1):19-25. doi: 10.1016/j.jpain.2006.05.010. Epub 2006 Nov 16. PMID 17113353
- [Background] Gronroos M, Pertovaara A. Capsaicin-induced central facilitation of a nociceptive flexion reflex in humans. Neurosci Lett. 1993 Sep 3;159(1-2):215-8. doi: 10.1016/0304-3940(93)90837-b. PMID 8264971
- [Background] LaMotte RH, Lundberg LE, Torebjork HE. Pain, hyperalgesia and activity in nociceptive C units in humans after intradermal injection of capsaicin. J Physiol. 1992 Mar;448:749-64. doi: 10.1113/jphysiol.1992.sp019068. PMID 1593488
- [Background] Qerama E, Fuglsang-Frederiksen A, Kasch H, Bach FW, Jensen TS. Effects of evoked pain on the electromyogram and compound muscle action potential of the brachial biceps muscle. Muscle Nerve. 2005 Jan;31(1):25-33. doi: 10.1002/mus.20182. PMID 15536622
- [Background] World Medical Association,
- [Background] WHO,
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Cavallone LF, Frey K, Montana MC, Joyal J, Regina KJ, Petersen KL, Gereau RW 4th. Reproducibility of the heat/capsaicin skin sensitization model in healthy volunteers. J Pain Res. 2013 Nov 7;6:771-84. doi: 10.2147/JPR.S53437. eCollection 2013. PMID 24232380
- [Background] Nawab SH, Chang SS, De Luca CJ. High-yield decomposition of surface EMG signals. Clin Neurophysiol. 2010 Oct;121(10):1602-15. doi: 10.1016/j.clinph.2009.11.092. Epub 2010 Apr 28. PMID 20430694
- [Background] Koh RG, Nachman AI, Zariffa J. Use of spatiotemporal templates for pathway discrimination in peripheral nerve recordings: a simulation study. J Neural Eng. 2017 Feb;14(1):016013. doi: 10.1088/1741-2552/14/1/016013. Epub 2016 Dec 21. PMID 28000616
- [Background] Martinez-Valdes E, Negro F, Laine CM, Falla D, Mayer F, Farina D. Tracking motor units longitudinally across experimental sessions with high-density surface electromyography. J Physiol. 2017 Mar 1;595(5):1479-1496. doi: 10.1113/JP273662. PMID 28032343
- [Background] Quiroga RQ, Nadasdy Z, Ben-Shaul Y. Unsupervised spike detection and sorting with wavelets and superparamagnetic clustering. Neural Comput. 2004 Aug;16(8):1661-87. doi: 10.1162/089976604774201631. PMID 15228749
- [Background] Ha SM, Kwon OY, Cynn HS, Lee WH, Kim SJ, Park KN. Selective activation of the infraspinatus muscle. J Athl Train. 2013 May-Jun;48(3):346-52. doi: 10.4085/1062-6050-48.2.18. Epub 2013 Feb 20. PMID 23675794
- [Background] Hoheisel U, Mense S, Simons DG, Yu XM. Appearance of new receptive fields in rat dorsal horn neurons following noxious stimulation of skeletal muscle: a model for referral of muscle pain? Neurosci Lett. 1993 Apr 16;153(1):9-12. doi: 10.1016/0304-3940(93)90064-r. PMID 8510831
- [Background] Arendt-Nielsen L, Graven-Nielsen T. Central sensitization in fibromyalgia and other musculoskeletal disorders. Curr Pain Headache Rep. 2003 Oct;7(5):355-61. doi: 10.1007/s11916-003-0034-0. PMID 12946288
- [Background] Graven-Nielsen T, Arendt-Nielsen L. Assessment of mechanisms in localized and widespread musculoskeletal pain. Nat Rev Rheumatol. 2010 Oct;6(10):599-606. doi: 10.1038/nrrheum.2010.107. Epub 2010 Jul 27. PMID 20664523
- [Background] Umeda M, Corbin LW, Maluf KS. Preliminary investigation of absent nociceptive flexion reflex responses among more symptomatic women with fibromyalgia syndrome. Rheumatol Int. 2013 Sep;33(9):2365-72. doi: 10.1007/s00296-013-2725-0. Epub 2013 Apr 4. PMID 23553516
- [Background] Ziegler EA, Magerl W, Meyer RA, Treede RD. Secondary hyperalgesia to punctate mechanical stimuli. Central sensitization to A-fibre nociceptor input. Brain. 1999 Dec;122 ( Pt 12):2245-57. doi: 10.1093/brain/122.12.2245. PMID 10581220
- [Background] Andersson JL, Lilja A, Hartvig P, Langstrom B, Gordh T, Handwerker H, Torebjork E. Somatotopic organization along the central sulcus, for pain localization in humans, as revealed by positron emission tomography. Exp Brain Res. 1997 Nov;117(2):192-9. doi: 10.1007/s002210050215. PMID 9419066
- [Background] Lim ECW, Sterling M, Stone A, Vicenzino B. Central hyperexcitability as measured with nociceptive flexor reflex threshold in chronic musculoskeletal pain: a systematic review. Pain. 2011 Aug;152(8):1811-1820. doi: 10.1016/j.pain.2011.03.033. Epub 2011 Apr 27. PMID 21524852
- [Background] Fernandez-Carnero J, Ge HY, Kimura Y, Fernandez-de-Las-Penas C, Arendt-Nielsen L. Increased spontaneous electrical activity at a latent myofascial trigger point after nociceptive stimulation of another latent trigger point. Clin J Pain. 2010 Feb;26(2):138-43. doi: 10.1097/AJP.0b013e3181bad736. PMID 20090441
- [Background] Stifani N. Motor neurons and the generation of spinal motor neuron diversity. Front Cell Neurosci. 2014 Oct 9;8:293. doi: 10.3389/fncel.2014.00293. eCollection 2014. PMID 25346659
- [Derived] Evans V, Koh RGL, Duarte FCK, Linde L, Amiri M, Kumbhare D. A randomized double blinded placebo controlled study to evaluate motor unit abnormalities after experimentally induced sensitization using capsaicin. Sci Rep. 2021 Jul 2;11(1):13793. doi: 10.1038/s41598-021-93188-7. PMID 34215800

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT04361149/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT04361149/ICF_001.pdf